CLINICAL TRIAL: NCT01495832
Title: Impact of Pulse-enriched Foods on Cognitive Function and Cardiometabolic Health in Obese Adults
Acronym: PULSA-2011
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of South Australia (Other)
Responsible Party: Principal Investigator, Dr. Peter Zahradka, Professor, Department of Physiology, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B2001:084
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: Adult Obesity; Cardiometabolic health; Pulse Foods; Beans, Peas, Lentils; Cognitive Function
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulse Group (Experimental): The pulse group will consume pulse-enriched foods designed to deliver ½ cup of pulses per day for 12 weeks.
  Interventions: Other: Pulse Group
- Control Group (Active Comparator): The control group will consume comparator foods for 12 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Pulse Group — The pulse group will consume pulse-enriched foods designed to deliver ½ cup of pulses per day for 12 weeks.
  Other Names: Sanitarium; Heinz; Simplot
  Arms: Pulse Group
Other: Control Group — The control group will consume comparator foods for 12 weeks.
  Arms: Control Group

SUMMARY:
The Canadian population, as is the case in most developed countries, is ageing and becoming increasingly overweight and/or obese. Both ageing and obesity are associated with reduced cognitive performance which can impact adversely on the ability to undertake daily activities and increases the risk of loss of independent living and reduced quality of life. The investigators predict that consumption of ½ cup of pulses per day for 12 weeks will improve cognitive function in older overweight/obese adults and thus decrease the rate of cognitive decline that occurs in this at-risk population.

DETAILED DESCRIPTION:
This is a multi-site, randomized, controlled, parallel, dietary intervention food study designed to examine the impact of pulse-enriched foods on cognitive function and cardiometabolic health in obese adults. Recruitment will consist of approximately 160 participants (n= 80 participants per site) at 2 sites located in Winnipeg and South Australia.

Participants will be randomly allocated to one of 2 groups; a pulse group or a control group. The pulse group will consume pulse-enriched foods designed to deliver ½ cup of pulses per day for 12 weeks. The control group will consume comparator foods for 12 weeks. The pulse and comparator food items will be provided to participants and they will be asked to incorporate these into their usual diet. Participants will be requested not to change their diet or physical activity habits during the study period, other than as required to comply with the study requirements. Five-day weighed food records will be completed during the week prior to baseline and during the final week of the study to monitor dietary intake, in particular intake of pulses. This will determine whether participants are incorporating the study foods as required, and will be used to evaluate associated changes in dietary intake and body weight, if they occur.

ELIGIBILITY:
Inclusion Criteria:

* Male or females, between 50-80 years of age
* Body Mass Index (BMI) of >25 kg/m2
* Must be on a stable regime for the past 6 months if taking medications or supplements for elevated lipids, blood pressure, glucose management, mood, pain, or insomnia
* Consume 1 or less servings of pulses per week
* Able to read and understand English
* Willing to comply with the protocol requirements
* Willing to provide informed consent.

Exclusion Criteria:

* Body weight ≥135 kg (since this exceeds the capability for Dual Energy X-ray Absorptiometry, i.e, DEXA scanning to assess body composition)
* Established cardiovascular, liver, or kidney disease
* Uncontrolled diabetes (hemoglobin HbA1c >8)
* A score of ≤23 on the Mini Mental State Examination
* Use of appetite suppressants or Orlistat (Xenical)
* Inability to consume pulse-enriched foods (i.e., beans, peas, chickpeas, and lentils) due to allergies or severe gastrointestinal reactions
* Pregnancy
* Smoking or only recently quit smoking (smoked any cigarettes within the last 12 months)
* Weight loss of ≥3kg of body weight within the 6 months prior to enrolling in the study
* Adherence to a weight loss diet or physical activity program designed to facilitate weight loss
* Acute or terminal illness.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Vascular Function | 12 weeks
  Vascular function will be assessed non-invasively (at baseline, Week 6, and Week 12) with measurement of arterial compliance (elasticity) by pulse wave analysis and pulse wave velocity. Measurement of arterial vasodilation will be done non-invasively to evaluate endothelial cells which line the blood vessels that regulate blood flow. Blood samples will be taken to assess markers of vascular function.
Cerebral Blood Flow Velocity (Australian Site only) | 12 Weeks
  Cerebral blood flow velocity will be assessed (baseline , Week 6, Week 12) by transcranial Doppler ultrasonography. This will serve as an index of arterial vasodilator responsiveness in the cerebral circulation. This will be performed by the Australian site only.

SECONDARY OUTCOMES:
Cognitive Function | 12 weeks
  A selection of cognitive tests will be administered (baseline, Week 6, and Week 12) by a qualified member of the study team to assess varying aspects of the participant's level of functioning cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zahradka, PhD, Principal Investigator — University of Manitoba
Locations (2):
- University of South Australia, Nutritional Psysiology Research Centre, Sansom Institute for Health, Adelaide, South Australia, Australia
- St. Boniface Hospital Research Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Katzmarzyk PT. The Canadian obesity epidemic, 1985-1998. CMAJ. 2002 Apr 16;166(8):1039-40. No abstract available. PMID 12002980
- [Background] Raine K. Overweight and obesity in Canada: a population health perspective. Alberta: Centre for Health Promotion Studies, University of Alberta, 2004.
- [Background] Cameron AJ, Welborn TA, Zimmet PZ, Dunstan DW, Owen N, Salmon J, Dalton M, Jolley D, Shaw JE. Overweight and obesity in Australia: the 1999-2000 Australian Diabetes, Obesity and Lifestyle Study (AusDiab). Med J Aust. 2003 May 5;178(9):427-32. doi: 10.5694/j.1326-5377.2004.tb05998.x. PMID 12720507
- [Background] Tjepkema M. Adult obesity in Canada: measured height and weight. Nutrition: Findings from the Canadian Community Health Survey. Ottawa, 2005.
- [Background] Australian Bureau of Statistics. National Health Survey 2007-2008. In: Australian Institute of Health and Welfare, ed. Canberra: Commonwealth of Australia, 2009.
- [Background] Poirier P, Giles TD, Bray GA, Hong Y, Stern JS, Pi-Sunyer FX, Eckel RH; American Heart Association; Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Obesity and cardiovascular disease: pathophysiology, evaluation, and effect of weight loss: an update of the 1997 American Heart Association Scientific Statement on Obesity and Heart Disease from the Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Circulation. 2006 Feb 14;113(6):898-918. doi: 10.1161/CIRCULATIONAHA.106.171016. Epub 2005 Dec 27. PMID 16380542
- [Background] Elias MF, Elias PK, Sullivan LM, Wolf PA, D'Agostino RB. Lower cognitive function in the presence of obesity and hypertension: the Framingham heart study. Int J Obes Relat Metab Disord. 2003 Feb;27(2):260-8. doi: 10.1038/sj.ijo.802225. PMID 12587008
- [Background] Elias MF, Elias PK, Sullivan LM, Wolf PA, D'Agostino RB. Obesity, diabetes and cognitive deficit: The Framingham Heart Study. Neurobiol Aging. 2005 Dec;26 Suppl 1:11-6. doi: 10.1016/j.neurobiolaging.2005.08.019. Epub 2005 Oct 11. PMID 16223549
- [Background] Kilander L, Nyman H, Boberg M, Lithell H. Cognitive function, vascular risk factors and education. A cross-sectional study based on a cohort of 70-year-old men. J Intern Med. 1997 Oct;242(4):313-21. doi: 10.1046/j.1365-2796.1997.00196.x. PMID 9366810
- [Background] Sorensen TI, Sonne-Holm S, Christensen U, Kreiner S. Reduced intellectual performance in extreme overweight. Hum Biol. 1982 Dec;54(4):765-75. No abstract available. PMID 7166298
- [Background] Health Canada and Interdepartmental Committee on Aging and Seniors Issues. Canada's Aging Population. In: Minister of Public Works and Government Services, ed.: Health Canada, 2002.
- [Background] Australian Bureau of Statistics. Population projections Australia 2001-2101. Canberra: Commonwealth of Australia, 2003.
- [Background] Lakatta EG, Levy D. Arterial and cardiac aging: major shareholders in cardiovascular disease enterprises: Part II: the aging heart in health: links to heart disease. Circulation. 2003 Jan 21;107(2):346-54. doi: 10.1161/01.cir.0000048893.62841.f7. No abstract available. PMID 12538439
- [Background] Versari D, Daghini E, Virdis A, Ghiadoni L, Taddei S. The ageing endothelium, cardiovascular risk and disease in man. Exp Physiol. 2009 Mar;94(3):317-21. doi: 10.1113/expphysiol.2008.043356. Epub 2008 Sep 19. PMID 18805864
- [Background] Guidelines for the evaluation of dementia and age-related cognitive decline. American Psychological Association Presidential Task Force. Am Psychol. 1998 Dec;53(12):1298-303. PMID 9872051
- [Background] Fjeldstad AS, Montgomery PS, Gardner AW. Age-related differences in arterial compliance are independent of body mass index. Angiology. 2008 Aug-Sep;59(4):454-8. doi: 10.1177/0003319707306455. Epub 2008 Apr 2. PMID 18388081
- [Background] Wildman RP, Mackey RH, Bostom A, Thompson T, Sutton-Tyrrell K. Measures of obesity are associated with vascular stiffness in young and older adults. Hypertension. 2003 Oct;42(4):468-73. doi: 10.1161/01.HYP.0000090360.78539.CD. Epub 2003 Sep 2. PMID 12953016
- [Background] Fujiwara Y, Chaves PH, Takahashi R, Amano H, Yoshida H, Kumagai S, Fujita K, Wang DG, Shinkai S. Arterial pulse wave velocity as a marker of poor cognitive function in an elderly community-dwelling population. J Gerontol A Biol Sci Med Sci. 2005 May;60(5):607-12. doi: 10.1093/gerona/60.5.607. PMID 15972613
- [Background] Hanon O, Haulon S, Lenoir H, Seux ML, Rigaud AS, Safar M, Girerd X, Forette F. Relationship between arterial stiffness and cognitive function in elderly subjects with complaints of memory loss. Stroke. 2005 Oct;36(10):2193-7. doi: 10.1161/01.STR.0000181771.82518.1c. Epub 2005 Sep 8. PMID 16151027
- [Background] Nagai K, Akishita M, Machida A, Sonohara K, Ohni M, Toba K. Correlation between pulse wave velocity and cognitive function in nonvascular dementia. J Am Geriatr Soc. 2004 Jun;52(6):1037-8. doi: 10.1111/j.1532-5415.2004.52277_15.x. No abstract available. PMID 15161489
- [Background] Scuteri A, Brancati AM, Gianni W, Assisi A, Volpe M. Arterial stiffness is an independent risk factor for cognitive impairment in the elderly: a pilot study. J Hypertens. 2005 Jun;23(6):1211-6. doi: 10.1097/01.hjh.0000170384.38708.b7. PMID 15894897
- [Background] Fukuhara M, Matsumura K, Ansai T, Takata Y, Sonoki K, Akifusa S, Wakisaka M, Hamasaki T, Fujisawa K, Yoshida A, Fujii K, Iida M, Takehara T. Prediction of cognitive function by arterial stiffness in the very elderly. Circ J. 2006 Jun;70(6):756-61. doi: 10.1253/circj.70.756. PMID 16723799
- [Background] Kim YS, Kim DH, Choi BH, Sohn EH, Lee AY. Relationship between brachial-ankle pulse wave velocity and cognitive function in an elderly community-dwelling population with metabolic syndrome. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):176-9. doi: 10.1016/j.archger.2008.07.004. Epub 2008 Sep 10. PMID 18786736
- [Background] Scuteri A, Tesauro M, Appolloni S, Preziosi F, Brancati AM, Volpe M. Arterial stiffness as an independent predictor of longitudinal changes in cognitive function in the older individual. J Hypertens. 2007 May;25(5):1035-40. doi: 10.1097/HJH.0b013e3280895b55. PMID 17414668
- [Background] Waldstein SR, Rice SC, Thayer JF, Najjar SS, Scuteri A, Zonderman AB. Pulse pressure and pulse wave velocity are related to cognitive decline in the Baltimore Longitudinal Study of Aging. Hypertension. 2008 Jan;51(1):99-104. doi: 10.1161/HYPERTENSIONAHA.107.093674. Epub 2007 Nov 19. PMID 18025297
- [Background] Anderson JW, Story L, Sieling B, Chen WJ, Petro MS, Story J. Hypocholesterolemic effects of oat-bran or bean intake for hypercholesterolemic men. Am J Clin Nutr. 1984 Dec;40(6):1146-55. doi: 10.1093/ajcn/40.6.1146. PMID 6095635
- [Background] Mathur KS, Khan MA, Sharma RD. Hypocholesterolaemic effect of Bengal gram: a long-term study in man. Br Med J. 1968 Jan 6;1(5583):30-1. doi: 10.1136/bmj.1.5583.30. No abstract available. PMID 5636741
- [Background] Anderson JW, Gustafson NJ, Spencer DB, Tietyen J, Bryant CA. Serum lipid response of hypercholesterolemic men to single and divided doses of canned beans. Am J Clin Nutr. 1990 Jun;51(6):1013-9. doi: 10.1093/ajcn/51.6.1013. PMID 2161614
- [Background] Duane WC. Effects of legume consumption on serum cholesterol, biliary lipids, and sterol metabolism in humans. J Lipid Res. 1997 Jun;38(6):1120-8. PMID 9215540
- [Background] Jenkins DJ, Wong GS, Patten R, Bird J, Hall M, Buckley GC, McGuire V, Reichert R, Little JA. Leguminous seeds in the dietary management of hyperlipidemia. Am J Clin Nutr. 1983 Oct;38(4):567-73. doi: 10.1093/ajcn/38.4.567. PMID 6624698
- [Background] Shutler SM, Bircher GM, Tredger JA, Morgan LM, Walker AF, Low AG. The effect of daily baked bean (Phaseolus vulgaris) consumption on the plasma lipid levels of young, normo-cholesterolaemic men. Br J Nutr. 1989 Mar;61(2):257-65. doi: 10.1079/bjn19890114. PMID 2650733
- [Background] Nagata C, Takatsuka N, Kurisu Y, Shimizu H. Decreased serum total cholesterol concentration is associated with high intake of soy products in Japanese men and women. J Nutr. 1998 Feb;128(2):209-13. doi: 10.1093/jn/128.2.209. PMID 9446845
- [Background] Anderson JW, Major AW. Pulses and lipaemia, short- and long-term effect: potential in the prevention of cardiovascular disease. Br J Nutr. 2002 Dec;88 Suppl 3:S263-71. doi: 10.1079/BJN2002716. PMID 12498626
- [Background] Bazzano LA, He J, Ogden LG, Loria C, Vupputuri S, Myers L, Whelton PK. Legume consumption and risk of coronary heart disease in US men and women: NHANES I Epidemiologic Follow-up Study. Arch Intern Med. 2001 Nov 26;161(21):2573-8. doi: 10.1001/archinte.161.21.2573. PMID 11718588
- [Background] Villegas R, Gao YT, Yang G, Li HL, Elasy TA, Zheng W, Shu XO. Legume and soy food intake and the incidence of type 2 diabetes in the Shanghai Women's Health Study. Am J Clin Nutr. 2008 Jan;87(1):162-7. doi: 10.1093/ajcn/87.1.162. PMID 18175751
- [Background] Feskens EJ, Virtanen SM, Rasanen L, Tuomilehto J, Stengard J, Pekkanen J, Nissinen A, Kromhout D. Dietary factors determining diabetes and impaired glucose tolerance. A 20-year follow-up of the Finnish and Dutch cohorts of the Seven Countries Study. Diabetes Care. 1995 Aug;18(8):1104-12. doi: 10.2337/diacare.18.8.1104. PMID 7587845
- [Background] Azadbakht L, Mirmiran P, Shiva N, Azizi F. General obesity and central adiposity in a representative sample of Tehranian adults: prevalence and determinants. Int J Vitam Nutr Res. 2005 Jul;75(4):297-304. doi: 10.1024/0300-9831.75.4.297. PMID 16229347
- [Background] Newby PK, Muller D, Hallfrisch J, Qiao N, Andres R, Tucker KL. Dietary patterns and changes in body mass index and waist circumference in adults. Am J Clin Nutr. 2003 Jun;77(6):1417-25. doi: 10.1093/ajcn/77.6.1417. PMID 12791618
- [Background] Schulz M, Kroke A, Liese AD, Hoffmann K, Bergmann MM, Boeing H. Food groups as predictors for short-term weight changes in men and women of the EPIC-Potsdam cohort. J Nutr. 2002 Jun;132(6):1335-40. doi: 10.1093/jn/132.6.1335. PMID 12042455
- [Background] Jimenez-Cruz A, Bacardi-Gascon M, Turnbull WH, Rosales-Garay P, Severino-Lugo I. A flexible, low-glycemic index mexican-style diet in overweight and obese subjects with type 2 diabetes improves metabolic parameters during a 6-week treatment period. Diabetes Care. 2003 Jul;26(7):1967-70. doi: 10.2337/diacare.26.7.1967. PMID 12832297
- [Background] Williams PG, Grafenauer SJ, O'Shea JE. Cereal grains, legumes, and weight management: a comprehensive review of the scientific evidence. Nutr Rev. 2008 Apr;66(4):171-82. doi: 10.1111/j.1753-4887.2008.00022.x. PMID 18366531
- [Background] Pittaway JK, Ahuja KD, Robertson IK, Ball MJ. Effects of a controlled diet supplemented with chickpeas on serum lipids, glucose tolerance, satiety and bowel function. J Am Coll Nutr. 2007 Aug;26(4):334-40. doi: 10.1080/07315724.2007.10719620. PMID 17906185
- [Background] Pittaway JK, Ahuja KD, Cehun M, Chronopoulos A, Robertson IK, Nestel PJ, Ball MJ. Dietary supplementation with chickpeas for at least 5 weeks results in small but significant reductions in serum total and low-density lipoprotein cholesterols in adult women and men. Ann Nutr Metab. 2006;50(6):512-8. doi: 10.1159/000098143. Epub 2006 Dec 21. PMID 17191025
- [Background] Nestel P, Cehun M, Chronopoulos A. Effects of long-term consumption and single meals of chickpeas on plasma glucose, insulin, and triacylglycerol concentrations. Am J Clin Nutr. 2004 Mar;79(3):390-5. doi: 10.1093/ajcn/79.3.390. PMID 14985212
- [Background] Pittaway JK, Robertson IK, Ball MJ. Chickpeas may influence fatty acid and fiber intake in an ad libitum diet, leading to small improvements in serum lipid profile and glycemic control. J Am Diet Assoc. 2008 Jun;108(6):1009-13. doi: 10.1016/j.jada.2008.03.009. PMID 18502235
- [Background] Zahradka, P., Guzman, R., Weighell, W., Wright, B., Baldwin, A., Louis, S., Rodriguez, D., and Taylor, C.G. 2009 Increased consumption of legumes improves arterial stiffness in peripheral vascular disease independent of blood pressure, weight and serum cholesterol. Experimental Biology 2009, April 18-22, New Orleans, LA. [oral presentation].
- [Background] Bouchard C, Tremblay A, Leblanc C, Lortie G, Savard R, Theriault G. A method to assess energy expenditure in children and adults. Am J Clin Nutr. 1983 Mar;37(3):461-7. doi: 10.1093/ajcn/37.3.461. PMID 6829488
- See also: St. Boniface General Hospital Research Centre — http://www.bing.com/search?q=st.+boniface+general+hospital+research+centre&form=DLCMHP&mkt=en-ca&qs=AS&sk=AS1&pq=st.+boniface+general+hospital&sp=2&sc=3-29
- See also: Canadian Centre for Agri-food Research in Health & Medicine — http://www4.agr.gc.ca/AAFC-AAC/display-afficher.do?id=1262627380265&lang=eng